CLINICAL TRIAL: NCT04162054
Title: Observation of Acute Cardiopulmonary Effects in Healthy Individuals Performing Cardiopulmonary Exercise Test (CPX) During Whole Body Vibration (WBV)
Acronym: GALILEOhealthy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Felix Gerhardt, Dr. med., Klinikum der Universität Köln
Other Study IDs: 003
Record Dates: First submitted 2019-04-25; First posted 2019-11-14 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Cardiopulmonary Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study to evaluate acute cardiopulmonary effects of whole body vibration (WBV) on healthy individuals analysed in non-invasive cardiopulmonary exercise test (CPX). — Observational study to evaluate acute cardiopulmonary effects of whole body vibration (WBV) on healthy individuals analysed in non-invasive cardiopulmonary exercise test (CPX).

SUMMARY:
Observational study to evaluate acute cardiopulmonary effects of oscillatory whole body vibration (WBV) on healthy individuals analysed in non-invasive cardiopulmonary exercise test (CPX).

DETAILED DESCRIPTION:
Oscillatory whole-body vibration (WBV) is a novel exercise modality, which is performed on a vibrating platform that moves in sinusoidal oscillations, and during which static and dynamic exercises can be performed. Rapid movements of the platform lead to muscle spindle reﬂexes, which result in reﬂectory contraction of muscle groups and thus promote gain of muscle strength and power. The most efﬁcient vibration rate enhancing muscle function is assumed to be ∼20 Hz, leading to constant muscle contraction and anaerobic metabolism of the affected muscle ﬁbres. As a consequence, lactate liberation serves as a stimulus for muscle gain.This methodology has been successfully utilised to enhance moving velocity, muscle power and strength in young athletes and chronic obstructive pulmonary disease though not been understood in all details. Therefore this investigation will help to evaluate acute cardiopulmonary effects of whole body vibration (WBV) on healthy individuals analysed in non-invasive cardiopulmonary exercise test (CPX).

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals planning on performing a WBV-Training
* healthy individuals planning on performing a CPX

Exclusion Criteria:

* exclusion to perform CPX
* exclusion to perform WBV

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * healthy individuals planning on performing a WBV-Training
  * healthy individuals planning on performing a CPX
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 in mililiter | one day
  maximal Oxygen saturation

SECONDARY OUTCOMES:
Nadir Co2 at anaerobic threshold | one day
  Nadir Co2 in mmHG
anaerobic threshold (AT) | one day
  AT in mililiter

CONTACTS AND LOCATIONS:
Locations (1):
- Spezialambulanz für pulmonale Hypertonie Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gerhardt F, Dumitrescu D, Gartner C, Beccard R, Viethen T, Kramer T, Baldus S, Hellmich M, Schonau E, Rosenkranz S. Oscillatory whole-body vibration improves exercise capacity and physical performance in pulmonary arterial hypertension: a randomised clinical study. Heart. 2017 Apr;103(8):592-598. doi: 10.1136/heartjnl-2016-309852. Epub 2017 Jan 18. PMID 28100544